CLINICAL TRIAL: NCT06791083
Title: Envafolimab Combined With Fruquintinib and Chemotherapy for Neoadjuvant Treatment of Gastric Cancer: a Single-arm, Open Clinical Study
Brief Title: Clinical Study of Envafolimab Combined With Fruquintinib and Chemotherapy for Neoadjuvant Treatment of Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-013-E1-GC003
Record Dates: First submitted 2024-06-20; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — envafolimab; HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Envafolimab combined with Fruquintinib and chemotherapy (Experimental)
  Interventions: Drug: Envafolimab; Drug: Fruquintinib

INTERVENTIONS:
Drug: Envafolimab — 150mg/m2 , IH， d1；Q3W
Drug: Fruquintinib — 5 mg ，po，QD，d1-d14；Q3W

SUMMARY:
To observe and evaluate the neoadjuvant treatment of Envafolimab combined with Fruquintinib and chemotherapy for locally advanced gastric/gastroesophageal junction carcinoma

DETAILED DESCRIPTION:
This study observed and evaluated the major pathological response rate (MPR), pathological complete response rate (pCR), pathological response rate (pRR), objective response rate (ORR), R0 removal rate, disease-free survival (DFS) of Envafolimab combined with Fruquintinib and chemotherapy in neoadjuvant therapy for locally advanced gastric/gastroesophageal junctional cancer. Overall survival (OS) and security. The relationship between tumor angiogenesis and lymphangiogenesis and clinical outcome of patients (including but not limited to immunohistochemical detection of CD31, CD3, CD8, etc.) was also explored.

ELIGIBILITY:
Inclusion Criteria:

1. Have fully understood the study and voluntarily signed the informed consent;
2. Aged 18-75 years (including 18 and 75 years);
3. Pathologically confirmed or potentially resectable locally advanced gastric/gastroesophageal junction adenocarcinoma (cT2-T4b, N+M0);
4. If bone metastasis is suspected, a bone scan should be performed. If peritoneal metastasis is suspected, abdominal examination should be performed to rule out distant metastasis.
5. At least 1 measurable lesion according to RECIST v1.1 criteria;
6. United States Eastern Cancer Consortium (ECOG) Physical status score 0-1; BMI≥18;
7. Expected survival ≥12 weeks;
8. The functions of vital organs during the first 14 days of enrollment met the following requirements:

   * Absolute neutrophil count ≥1.5×109/L;
   * Platelet ≥80×109/L;
   * Hemoglobin ≥90g/L;
   * Total bilirubin < 1.5 ULN; ALT and AST < 2.5 ULN (< 5 ULN in patients with liver metastasis);
   * Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (CCr)≥60ml/min;
   * endogenous creatinine clearance > 50ml/min;
9. Female subjects of childbearing age or male subjects whose sexual partner is a female of childbearing age should take effective contraceptive measures during the whole treatment period and 6 months after the treatment period;
10. Good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Known HER2-positive patients;
2. Participated in other drug clinical trials and received at least one drug therapy within 4 weeks prior to enrollment or received other systemic anti-tumor therapy, including chemotherapy, signal transduction inhibitors, immunotherapy, and other investigational drugs within 4 weeks prior to enrollment;
3. Had other malignancies within 5 years prior to admission, except basal cell or squamous cell carcinoma of the skin after radical surgery, or carcinoma in situ of the cervix;
4. Receive live vaccine within 4 weeks prior to enrollment or possibly during the study period;
5. Had active autoimmune disease or history of autoimmune disease within 4 weeks prior to enrollment;
6. Previously received allogeneic bone marrow transplantation or organ transplantation;
7. The patient has a current disease or condition that affects drug absorption, or the patient cannot take Fruquintinib orally;
8. Subjects who are allergic to the investigational drug or any of its adjuncts;
9. The investigator identified clinically significant electrolyte abnormalities;
10. Hypertension that could not be controlled by drugs before enrollment was defined as: systolic blood pressure ≥150 mmHg and/or diastolic blood pressure ≥100 mmHg;
11. Gastrointestinal diseases such as active ulcer of stomach and duodenum, ulcerative colitis, or active bleeding of unresectable tumors, or other conditions that may cause gastrointestinal bleeding or perforation as determined by researchers before enrollment;
12. Patients with significant evidence or history of bleeding tendency within 3 months (bleeding >30 mL within 3 months, accompanied by hematemesis, stool, and blood in the stool), hemoptysis (>5 mL of fresh blood within 4 weeks), or thromboembolic events (including stroke events and/or transient ischemic attacks) within 12 months prior to admission;
13. History of severe cardiovascular and cerebrovascular diseases:

    * Cerebrovascular accident (excluding lacunar infarction, minor cerebral ischemia, or transient ischemic attack), myocardial infarction, unstable angina, and poorly controlled arrhythmias (including QTc interval ≥ 450ms for men and 470 ms for women) within 6 months prior to first administration of the study drug (QTc interval Fridericia) Formula calculation);
    * New York Heart Association (NYHA) heart function Grade > II or left ventricular ejection fraction (LVEF) < 50%;
14. Known human immunodeficiency virus (HIV) infection; A known history of clinically significant liver disease, including viral hepatitis [active HBV infection, i.e., positive HBV DNA (>1×104 copies /mL or >2000 IU/ml) must be excluded for a known hepatitis B virus (HBV) carrier; Known hepatitis C virus infection (HCV) and HCV RNA positive (>1×103 copies /mL), or other hepatitis, cirrhosis];

16. Women who are pregnant (positive pregnancy test before medication) or breastfeeding; 17. Two consecutive routine urine tests indicated urine protein ≥2+, and the urine protein volume >1.0g within 24 hours of reexamination; 18. Patients with ascites or pleural effusion with clinical symptoms; 19. CTCAE V5.0 grade 1 or higher toxicity due to any previous anticancer treatment that is not resolved, excluding oxaliplatin induced alopecia, lymphocytopenia, and neurotoxicity ≤ grade 2; 20.Patients considered inappropriate for inclusion in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Major pathological response rate (MPR) | up to 12 months
  MPR is defined as the proportion of neoadjuvant therapy induced tumor regression with pathologically remaining tumor < 10%

SECONDARY OUTCOMES:
Pathological complete response rate (pCR) | up to 12 months
  pCR is defined as the proportion of patients who do not have residual cancer cells on pathological examination after treatment
Pathological response rate (pRR) | up to 12 months
  pRR is defined as the proportion of patients whose pathologic examination after treatment found no cancer cells remaining or whose cancer cells remaining within a pre-specified value range
Objective response rate (ORR) | up to 12 months
  ORR is defined as the proportion of patients whose best overall assessment is a complete or partial response.
Disease-free survival (DFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 years
  DFS is defined as the time between a patient's enrollment and the onset of tumor recurrence or death from any cause
Overall survival (OS) | From date of randomization until the date of death from any cause, assessed up to 10 years
  OS is defined as the time until a patient is enrolled and dies from any cause
R0 removal rate | up to 24 weeks
  R0 resection rate was defined as the proportion of patients with complete resection of the tumor and a negative submicroscopic margin, i.e. no residual tumor

OTHER OUTCOMES:
Relationship between tumor angiogenesis and lymphangiogenesis and clinical outcomes | Through study completion, an average of 1 year
  Investigate the relationship between tumor angiogenesis, lymphangiogenesis (including but not limited to immunohistochemical detection of CD31, CD3, CD8, etc. expression) and the clinical outcomes (PFS, OS, ORR, etc.) of patients

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No